CLINICAL TRIAL: NCT04200521
Title: The Effect of Bariatric Procedures on Gut Microbiota, Gut Peptide and Metabolism in Obese Individuals in United Arab Emirates and Lebanon
Brief Title: The Effect of Bariatric Procedures on Gut Microbiota in Obese Individuals in United Arab Emirates and Lebanon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zayed University (Other)
Responsible Party: Principal Investigator, Mirey Karavetian, Assistant Professor, Zayed University
Other Study IDs: 1234
Record Dates: First submitted 2019-07-11; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Bariatric Surgery; Microbiota; Obesity; Dysbiosis
Keywords: Gut peptide; Energy metabolism; Appetite
MeSH Terms: conditions — Obesity; Dysbiosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Stool microbiota analysis (stool analysis): for healthy and for obese participants (pre and post bariatric intervention after 3 months). Using Polymerase Chain Reaction products of the V3-V4 region of 16S rRNA gene will be sequenced using a barcoded Illumina paired-end sequencing technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy weight individuals: Cross-sectional observation on healthy participants who will be recruited from the general population from both genders (Lebanese and Emirati Subjects).
- Obese individuals: Prospective study of 3 months duration (pre and post design) on obese Emirati and Lebanese participants undergoing bariatric procedure irrelevant of the study, from Qassimi Hospital In sharja and Middle East Institute of Health University Hospital, Lebanon

SUMMARY:
Overweight and obesity are worldwide health problems that can affect negatively quality of life. With increasing prevalence of obesity and the failure of compliance to lifestyle, bariatric surgeries have become the treatment of choice to help achieve long term sustainable weight loss. In some cases of bariatric surgery, weight loss stops and there are cases in which obesity manifests itself again; the mechanism underlying the re-appearance of obesity is not known. Recently, the gut microbiota, has been implicated in the etiology of obesity and metabolic syndrome due to its important role in digestion, metabolism and regulating gut peptides and hormones. In accordance with this, it has been shown in mice that obesity can be associated with dysbiosis (Imbalance in gut bacteria) and there has been successful reduction of weight in interventions when microbiota was manipulated.

Hypothesis:

1. Emirati participants will have unique microbiota and gut peptides when compared to Lebanese participants.
2. The microbiota and gut peptides variability is significantly different between those with normal weight compared to obese participants undergoing bariatric surgery.
3. The bariatric procedure will have a significant effect on the variability of microbiota, gut peptides, blood chemistry, dietary intake and metabolism among the obese participants.

Objectives of the study:

1. Determine the gut microbiota composition of Emirati healthy normal weight participants and compare to that of Lebanese via Illumina sequencing NGS (Next Generation Sequencing of the 16S rRNA gene) of the microbiota from the stool samples.
2. Determine the gut microbiota composition of Emirati obese participants and compare to that of Lebanese counterparts using NGS.
3. Determine the effect of bariatric procedure in UAE and Lebanon respectively on gut microbiota (using NGS), gut peptides in plasma, blood chemistry and metabolism using indirect calorimetry and food intake.

Importance of this research:

The microbiota and gut peptides variability is determined by body weight and ethnicity of the studied populations. It is hypothesized that bariatric surgery will have a significant effect on the variability of microbiota, gut peptides, blood chemistry, dietary intake and metabolism. This study will be a pioneering research in UAE and Lebanon to assist in finding population tailored therapeutic strategies that target the gut microbiota and treat obesity.

DETAILED DESCRIPTION:
This study has two arms: 1) cross-sectional observation on healthy participants, and 2) multi-center, prospective study of 3 month duration (pre and post design) on obese participants undergoing bariatric procedure.

Population study: Forty Emirati obese adults from UAE and 40 Lebanese obese adults from Lebanon from both genders and planning to undergo bariatric procedure (irrelevant of the study) will be recruited. All participants planning to conduct the surgery will be contacted; the consenting ones will be recruited till target sample saturation. Afterwards, 40 healthy counterparts from each country will be selected. Healthy participants will be recruited from Zayed University or staff of Qassimi Hospital in Sharjah, UAE and from staff/students/colleagues of the Middle East Institute of Health University Hopsital in Lebanon.

Assessment and Data Collection: 2 Research assistants (one in each hospital) will be trained by the principal investigator (PI) on the study instruments and data collection methods. These assistants will administer 4 questionnaires for each participant (healthy and obese per-operatively) at baseline(t0) and 4 questionnaires for the obese participants after the bariatric procedure after 3 months (t1). For quality control purposes, each questionnaire will be administered to all patients before the administration of the following questionnaire. Furthermore, each questionnaire will be completed and reviewed prior to administering the next. The assessment will take place in the specified clinic or hospital.

All of the parameters, except the demographics and initial screening questionnaire (collected only at t0) and follow up post bariatric questionnaire (t1: at 3 months, after the bariatric procedure), will be collected and monitored at 2 time points: Baseline (t0: at the beginning of the study), and follow up for obese participants (t1: at 3 months, after the bariatric procedure).

Assessment tools include:

Demographics

Questionnaires for:

i. Initial screening questionnaire ii. Follow up post bariatric questionnaire iii. 24 hour recall iv. Anxiety and Stress Levels using the DASS v. Appetite questionnaire

All questionnaires that are originally not in Arabic, will be translated to Arabic (local language), prior to study by translators whose first language is Arabic and back translated to English to assure coherence with original version.

Biochemical evaluation

An overnight fast of at least 12 h for blood collection is required. Collection will be done by a certified nurse at the Middle East institute of Health University Hospital and Qassimi Hospital. The blood will be analyzed for the following parameters:

* Lipid and glucose profile: serum triglyceride, total cholesterol, HDL-cholesterol, LDL- cholesterol, fasting blood glucose,
* Gut peptides: Total GLP-1, GLP-2, PYY, CCK, Ghrelin,
* Hormones: fasting insulin and Leptin

The questionnaires will be administered during the participants' routine visits. And blood draw will be taken during that visit (for obese participants,around 1 week prior to surgery) And 3 months post bariatric surgery for obese individuals. For each time, for the complete process, a total of 30 min will be needed per participant.

Nutritional Assessment • Anthropometric measurements will be assessed through a dietitian at the Middle East institute of Health University Hospital in Lebanon and Qassimi Hospital in sharjah, UAE. It will include body weight, body height, Body mass index (BMI), waist circumference (WC). Body composition will be evaluated using bioelectrical impedance analysis and energy expenditure using portable Indirect Calorimeter.

Fecal microbiota analysis.

• Participants will be given special collection kits followed by instructions on how to collect the stool. They will be asked to inform the research team when the samples are ready, so it will be collected within 24 hours. 2 samples will be collected from each participant, where 1 will be analyzed and second kept for accuracy check. Stool microbiota analysis will be done for all the participants at baseline and repeated at 3 months for the obese participants post bariatric surgery. Using Polymerase Chain Reaction (PCR) products of the V3-V4 region of 16S rRNA gene will be sequenced using a barcoded Illumina paired-end sequencing technique. The primary composition of the microbiome in the stool samples will be determined and analyzed by cluster analysis.

Sample size was determined according to change in Bacteroidetes/Firmicutes ratio, considering it as the main objective outcome of this study. Calculations were based on the data retrieved from Damms-Machado et al (2015) where serum Bacteroidetes/Firmicutes ratio changed significantly from 5.9 ±2.1 to 10.4± 1.4 in 3 months post bariatric surgery.To generate a similar significant effect of a sample size of 2 participants was estimated to achieve 80% power at a 5% alpha. Expecting a drop in effect size in this protocol, a high attrition rate among the samples at 3 months; we multiplied the number of participants in it by 20. Thus a sample of 40 participants per groups was planned for this study.

Data will be analyzed through SPSS version 18. Correlations will be conducted through ANOVA. Effect of the study will be analyzed by paired t test on continuous data and Chi square on categorical data. Microbiota composition will be analyzed using QIIME, and alpha- and beta-diversity will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Emirati residing in UAE and Lebanese residing in Lebanon
* 18 to 60 years old - from both genders
* Free of antibiotics for at least 3 months
* Two BMI categories: 1) obese with a BMI of ≥35 kg/m2 planning to undergo a bariatric procedure 2) healthy counterparts with a BMI of 18.5-24.9 kg/m2

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria
* Consumption of alcohol above the recommended amount per day (>½ ounce of ethanol for females and >1 ounce for men)
* Pregnant at the time of the study
* Significant voluntary weight loss (≥5% in the preceding 3 months)
* Not willing to provide written consent to the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty Emirati obese adults from UAE and 40 Lebanese obese adults from Lebanon from both genders and planning to undergo bariatric procedure (irrelevant of the study) will be recruited. All participants planning to conduct the surgery will be contacted, the consenting ones will be recruited till target sample saturation. Afterwards, 40 healthy counterparts from each country will be selected. Healthy participants can be employees from Qassimi HospitaI in sharjah and Middle East Institute of Health University Hopsital in Lebanon or any healthy Emirati and Lebanese people willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-10-27 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut Microbiota composition in obese participants | Baseline and 3 months post bariatric surgery
  Using Illumina sequencing NGS (Next Generation Sequencing of the 16S rRNA gene) of the microbiota from the stool samples.

SECONDARY OUTCOMES:
Changes in plasma level of CCK Hormone in obese participants | Baseline and 3 months post bariatric surgery
  Via Blood test
Changes in plasma level of PYY Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of Ghrelin Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of Leptin Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of Insulin Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of GLP1 Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of GLP2 Hormone in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of fasting Cholesterol in obese participants | Baseline and 3 month post bariatric surgery
  Via Blood test
Changes in plasma level of Fasting Blood Sugar in obese participants | Baseline and 3 month post bariatric surgery
  Using Blood test
Assessing changes in Energy Expenditure in obese participants | Baseline and 3 months post bariatric surgery
  By using Indirect Calorimeter
Assessing changes in appetite in obese participants | Baseline and 3 months post bariatric surgery
  Using Simplified Nutritional Appetite Questionnaire. Following numerical scale: a =1, b =2, c = 3, d =4, e = 5. The sum of the scores for the individual items constitutes the SNAQ score. SNAQ score 14 indicates significant risk of at least 5% weight loss within six months.
Changes in Dietary Intake in obese participants | Baseline and 3 months post bariatric surgery
  Using 24 Hour dietary recall method. The method consists of precisely recalling, describing and quantifying the intake of foods and beverages consumed in the 24 hour period.
Measure the changes in emotional states of Depression, Anxiety and Stress.in obese participants | Baseline and 3 months post bariatric surgery
  Using Depression, Anxiety and Stress Scale - 21 Items (DASS-21) Each of the three DASS scales contains 14 items, divided into subscales of 2-5 items with similar content. Subjects are asked to use 4-point severity/frequency scales to rate the extent to which they have experienced each state over the past week. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items.
Changes in Body Composition in obese participants | Baseline and 3 months post bariatric surgery
  Via Bio-electrical Impedance Analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mirey Karavetian, PhD, Principal Investigator — Zayed University
Locations (2):
- Middle East Institute of Health, University Hospital, Beirut, Lebanon
- Al Qassimi Hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lovibond, S.H. & Lovibond, P.F. Manual for the Depression Anxiety & Stress Scales. (2nd Ed.)Sydney. Psychology Foundation 1995.
- [Background] Damms-Machado A, Mitra S, Schollenberger AE, Kramer KM, Meile T, Konigsrainer A, Huson DH, Bischoff SC. Effects of surgical and dietary weight loss therapy for obesity on gut microbiota composition and nutrient absorption. Biomed Res Int. 2015;2015:806248. doi: 10.1155/2015/806248. Epub 2015 Feb 1. PMID 25710027
- [Result] Cannon CP, Kumar A. Treatment of overweight and obesity: lifestyle, pharmacologic, and surgical options. Clin Cornerstone. 2009;9(4):55-68; discussion 69-71. doi: 10.1016/s1098-3597(09)80005-7. PMID 19789064
- [Result] Seganfredo FB, Blume CA, Moehlecke M, Giongo A, Casagrande DS, Spolidoro JVN, Padoin AV, Schaan BD, Mottin CC. Weight-loss interventions and gut microbiota changes in overweight and obese patients: a systematic review. Obes Rev. 2017 Aug;18(8):832-851. doi: 10.1111/obr.12541. Epub 2017 May 19. PMID 28524627
- [Result] Aydin S. Can Peptides and Gut Microbiota Be Involved in the Etiopathology of Obesity? Obes Surg. 2017 Jan;27(1):202-204. doi: 10.1007/s11695-016-2429-0. No abstract available. PMID 27787759
- [Result] Bauer PV, Hamr SC, Duca FA. Regulation of energy balance by a gut-brain axis and involvement of the gut microbiota. Cell Mol Life Sci. 2016 Feb;73(4):737-55. doi: 10.1007/s00018-015-2083-z. Epub 2015 Nov 5. PMID 26542800
- [Result] Cani PD, Osto M, Geurts L, Everard A. Involvement of gut microbiota in the development of low-grade inflammation and type 2 diabetes associated with obesity. Gut Microbes. 2012 Jul-Aug;3(4):279-88. doi: 10.4161/gmic.19625. Epub 2012 May 14. PMID 22572877
- [Result] Corfe BM, Harden CJ, Bull M, Garaiova I. The multifactorial interplay of diet, the microbiome and appetite control: current knowledge and future challenges. Proc Nutr Soc. 2015 Aug;74(3):235-44. doi: 10.1017/S0029665114001670. Epub 2015 Jan 23. PMID 25612669
- [Result] Patrone V, Vajana E, Minuti A, Callegari ML, Federico A, Loguercio C, Dallio M, Tolone S, Docimo L, Morelli L. Postoperative Changes in Fecal Bacterial Communities and Fermentation Products in Obese Patients Undergoing Bilio-Intestinal Bypass. Front Microbiol. 2016 Feb 23;7:200. doi: 10.3389/fmicb.2016.00200. eCollection 2016. PMID 26941724
- [Result] Round JL, Mazmanian SK. The gut microbiota shapes intestinal immune responses during health and disease. Nat Rev Immunol. 2009 May;9(5):313-23. doi: 10.1038/nri2515. PMID 19343057
- [Result] Adlerberth I, Wold AE. Establishment of the gut microbiota in Western infants. Acta Paediatr. 2009 Feb;98(2):229-38. doi: 10.1111/j.1651-2227.2008.01060.x. PMID 19143664
- [Result] Wilson MM, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr. 2005 Nov;82(5):1074-81. doi: 10.1093/ajcn/82.5.1074. PMID 16280441